CLINICAL TRIAL: NCT06825572
Title: Mesenchymal Stem Cells-Derived Extracellular Vesicles (MSC-EV) in Acute/Acute-on-Chronic Liver Failure After Liver Transplantationa：a Prospective, Randomized, Controlled Clinical Study
Brief Title: MSC-EVs in Acute/ Acute-on-Chronic Liver Failure After Liver Transplantation
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jun Zheng, Doctor of Department of Hepatic Surgery and Liver Transplantation Center of the Third Affiliated Hospital, Organ Transplantation Institute, Sun Yat-sen University, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC-EVs of ThirdSunYatSen
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Liver Failure; Mesenchymal Stem Cell; Extracellular Vesicles
Keywords: MSC-EV; Liver transplantation; Liver failure
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MSC-EVs group (Experimental): After liver transplantation, on the basis of postoperative standard treatment (anti-infection treatment, immunosuppressive treatment, nutritional support treatment, etc.), an additional injection of MSC-EV will be received between the 1st and 5th days after transplantation
  Interventions: Biological: MSC-EVs
- Non-MSC-EVs group (No Intervention): After liver transplantation, patients will receive postoperative standard treatment (anti-infection treatment, immunosuppressive treatment, nutritional support treatment, etc.)

INTERVENTIONS:
Biological: MSC-EVs — 10 E10 MSC-EV particles per 100ml for a single dose. No prior HLA matching between MSC donors and recipients or liver donors
  Arms: MSC-EVs group

SUMMARY:
Acute liver failure (ALF) refers to a potentially reversible disorder that was the result of severe liver injury, with an onset of encephalopathy within 8 weeks of symptom appearance and in the absence of pre-existing liver disease. Acute-on-chronic liver failure refers to a liver failure syndrome in which some patients with chronic liver disease with relatively stable liver function suffer from acute liver decompensation and liver failure due to the effects of various acute injury factors. Liver transplantation is the only curative treatment for this type of end-stage liver disease. The potential of MSCs to repair or regenerate damaged tissue and suppress immune responses makes them promising in the treatment of liver diseases, especially in the field of liver transplantation. Many studies have shown that MSC-based therapies can reduce the symptoms of liver disease due to their paracrine effects. Therefore, compared to the cells they derive from, mesenchymal stem cells-derived extracellular vesicles (MSC-EV) are gradually gaining attention for their enhanced safety, as they do not replicate or cause microvascular embolism, and can be easily stored without losing their properties. It represents a novel and effective cell-free therapeutic agent as alternative to cell-based therapies for liver diseases, and liver failure was also concerned. This study was designed to evaluate the safety and tolerability of MSC-EV in acute-on-chronic liver failure after liver transplantation.

DETAILED DESCRIPTION:
In the MSC-EV group (experimental group), 15 patients will receive a single injection of MSC-EV after their first liver transplantation. In the non-MSC-EV group (control group), 15 patients will not receive MSC-EV therapy after their first liver transplantation.

The outcome of the experimental group will be compared with that of similar control patients undergoing liver transplantation but who will not receive MSC-EV. Both of the two groups will receive standard immunosuppressive therapy( a regimen based on tacrolimus (TAC), mycophenolate mofetyl (MMF) and steroids). Patients participated in the experimental cohort will be infused with a single dose of 10 E10 MSC-EV particles per 100ml, at an appropriate time during the first 1-5 days after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70 years;
* Acute on chronic liver failure-which is characterized by acute hepatic insult manifesting as jaundice (serum total bilirubin [TBil] ≥ 10×ULN umol/L) and coagulopathy (international normalized ratio [INR] ≥ 1.5 or prothrombin activity < 40%), complicated within 4 weeks by ascites and/or encephalopathy as determined by physical examination, in patients with previously diagnosed or undiagnosed chronic liver disease; Requiring liver transplantation due to acute on chronic liver failure;
* Obtain the patients' consent after informing patients of the purpose and method of the clinical trial;

Exclusion Criteria:

* Past history of malignant disease
* Active uncontrolled infection;
* Combined transplantation
* EBV-negative;
* HIV or HCV positive;
* Retransplantation;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with MSC-EV infusion-related toxicity as assessed by CTCAE v4.0. | 24 hours after injection
  Incidence, timing and severity of any clinical complication related to MSC-EV infusion, such as tympanic body temperature, heart rate, mean arterial blood pressure and allergy, as assessed by CTCAE v4.0 .
Aspartate aminotransferase (AST) | 6 months after transplantation
  Collect clinical results reflecting liver function
Alanine aminotransferase (ALT) | 6 months after transplantation
  Collect clinical results reflecting liver function
Bilirubin level | 6 months after transplantation
  Collect clinical results reflecting liver function
International normalized ratio (INR) | 6 months after transplantation
  Collect clinical results reflecting liver function
carbohydrate Compound antigen (GGT) level | 6 months after transplantation
  Collect clinical results reflecting liver function
Adverse events | 6 months after transplantation
  Any adverse events which may related to MSC-EV infusion

SECONDARY OUTCOMES:
Number of survived patients at 1 year after liver transplantation, according to the follow-up results. | 12 months
  Patients who are surviving, as assessed by outpatient or telephone follow-up, at 1 year after liver transplantation
Number of survived grafts at 1 year after liver transplantation, according to the follow-up results. | 12 months
  Surviving patients with primary and functional grafts, as assessed by outpatient or telephone follow-up, at 1 year after liver transplantation.
Recipient's immune function, as assessed by analysis of immune cell subsets from biopsy or blood samples ,at months 1-6 after liver transplantation. | 6 months after transplantation
  A series of immune cell subsets will be analyzed, including T cells (CD3+), CD4+ T cells (CD3+ CD4+ lymphocytes), CD8+ T cells (CD3+ CD8+ lymphocytes), naïve CD4+ T cells (CD4+ CD45RAhigh lymphocytes), memory CD4+ T cells (CD4+ CD45RO+ lymphocytes), natural killer (NK) cells (CD3- CD56+ lymphocytes), as well as B cells (CD19+ lymphocytes)

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yang, PHD, MD, Study Director — Third Affiliated Hospital, Sun Yat-Sen University, guangzhou, Guangdong, China
Locations (1):
- Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China